CLINICAL TRIAL: NCT02344303
Title: A Single-dose, Open-label, Fixed Sequence, Two Period Cross Over Study to Assess the Tolerability of a Supra Therapeutic Dose of TRV130 Followed by A Single Dose, Randomized, Double Blind, Comparative, Positive and Placebo Controlled, Four Period Cross-over Study of the Effects of TRV130, at Therapeutic and Supra Therapeutic Doses, on the QTc Intervals in Healthy Subjects
Brief Title: Study of the Effects of TRV130, at Therapeutic and Supra Therapeutic Doses, on QTc Intervals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CP130-1008
Record Dates: First submitted 2015-01-09; First posted 2015-01-22 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Healthy
MeSH Terms: interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Fixed sequence, open label
  Interventions: Drug: TRV130
- Part B (Experimental): 4 way cross over, double blind
  Interventions: Drug: TRV130; Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: TRV130
Drug: Moxifloxacin
  Arms: Part B
Drug: Placebo
  Arms: Part B

SUMMARY:
Assess the electrocardiogram effects of TRV130 relative to placebo at therapeutic and supratherapeutic doses.

DETAILED DESCRIPTION:
* Part A of the study will assess clinical safety data of TRV130
* Part B of the study will assess the effect of single dose TRV130 on QTc

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 45 inclusive.
* Women must be either a) post-menopausal; b) surgically sterile; c) of child-bearing potential and practicing contraception or remaining sexually inactive.
* Men must be willing to abstain from sperm donation from the time of Screening through the Follow-up Visit and, if sexually active with a woman of child-bearing potential, must be protected by acceptable forms of effective contraception through the Follow-up Visit.

Exclusion Criteria:

* Past or present diseases including, but not limited to, significant medical abnormalities including: psychiatric, neurologic, pulmonary, cardiac, gastrointestinal, genitourinary, renal, metabolic, endocrinologic or autoimmune disorders.
* Has previously participated in another TRV130 clinical study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Part A - Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Prior to dose through 4 hours
Part B - Change from baseline in QTc | Prior to dose through 24 hours

SECONDARY OUTCOMES:
Part B - Pharmacodynamics - QTc | Prior to dose through 24 hours
  Including QTc, heart rate, PR interval, QRS interval, uncorrected QT interval, ECG morphology and correlation between the QTcF change from baseline and plasma concentrations of TRV130.
Part B - Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Prior to dose through Follow-Up Visit
  Adverse events reporting, clinical observations, 12- lead electrocardiograms, vital signs, respiratory rate, body temperature and safety laboratory tests
Part A & B - Pharmacokinetics - Cmax, tmax, AUC | Prior to dose through 24 hours
  Parameters will include (but not limited to): Cmax, tmax, AUC0-τ, z: (apparent terminal rate constant calculated from the regression analysis (slope) of the log-transformed measured concentrations on the terminal phase of the time)

CONTACTS AND LOCATIONS:
Overall Officials: Franck Skobieranda, Study Director — Trevena Inc.
Locations (1):
- Baltimore, Maryland, United States